CLINICAL TRIAL: NCT06087718
Title: Introduction of the Maastro Applicator for Endoluminal Boosting in Rectal Cancer: a Pilot Study
Brief Title: Feasibility of the Maastro Applicator in Rectal Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Feasibility Maastro applicator
Record Dates: First submitted 2023-09-27; First posted 2023-10-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer; Feasibility; Toxicity; Quality of Life; Radiation Toxicity; Radiation Proctitis; Brachytherapy; Complete Response
MeSH Terms: conditions — Rectal Neoplasms; Radiation Injuries; Pathologic Complete Response

STUDY DESIGN:
Intervention Model Description: A single arm prospective interventional pilot trial in 10 patients with feasibility and safety checks and early stopping/intermission rules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Maastro applicator in combination with chemoradiotherapy (Experimental): The intervention is similar to the treatment of arm B of the published OPERA trial, however the endoluminal boost will be given using the Maastro applicator instead of a CXRT device.
  Interventions: Device: Maastro applicator

INTERVENTIONS:
Device: Maastro applicator — The dose profile of the Maastro applicator is similar to the dose profile of a CXRT device. Patients will be stratified based on tumor size. The cut-off is set at the maximum diameter of the treatment surface of the Maastro applicator. The boost consists of 3 fractions with a dose equivalent to 30 Gy per fraction prescribed at the surface of the applicator. The 3 boost fractions will be delivered over a 4-week time period. Patients with a tumor size < 2.5 cm will receive an upfront boost followed by concurrent chemoradiotherapy (25x1.8 Gy combined with capecitabine 825 mg/m2 bd on radiotherapy days). Patients with a tumor size ≥ 2.5cm will first undergo concurrent chemoradiotherapy (25x1.8 Gy combined with capecitabine 825 mg/m2 bd on radiotherapy days) and will afterwards receive the boost.

SUMMARY:
The goal of this interventional pilot trial is to confirm that Maastro endoluminal HDR ( High Dose Radiation) contact brachytherapy boosting is feasible and may increase the chance of functional organ sparing of the rectum in patients with rectal cancer. Participants will be treated with chemoradiotherapy and an endoluminal boost with the Maastro applicator.

DETAILED DESCRIPTION:
The goal of this clinical trial is to confirm that Maastro endoluminal HDR contact brachytherapy boosting is feasible and may increase the chance of functional organ sparing of the rectum in patients with rectal cancer. If at least 7 out of 10 planned Maastro applicator treatment series (3 fractions per series) can be conducted successfully from a procedural point of view the treatment will be considered feasible. The study intervention will be similar to the study treatment of arm B of the OPERA trial. Opposed to the treatment in arm B of the OPERA trial, the endoluminal boost will be given using HDR brachytherapy with the Maastro applicator instead of a CXRT (Contact X-ray Radiotherapy) device. The dose profile of the Maastro applicator is similar to the dose profile of CXRT device. As in the OPERA trial patients will be stratified based on tumor size. As the diameter of the treatment field of the largest Maastro applicator (there are two sizes) equals 2.5 cm we will stratify for tumor diameter < 2.5 cm v ≥ 2.5 cm. In the OPERA trial patients were stratified for a tumor diameter of < 3.0 cm v ≥ 3.0 cm as currently the largest applicator diameter for the CXRT device is 3.0 cm (currently available applicators: 2.0, 2.5 and 3.0 cm). The endoluminal boost will consist of 3 fractions with a dose equivalent to 30 Gy per fraction prescribed at the surface of the applicator. The 3 boost fractions will be delivered over a 4-week time period (week 1-2-4). Conform OPERA protocol, patients with a tumor size < 2.5 cm will receive an upfront endoluminal HDR contact boost followed by concurrent chemoradiotherapy (25x1.8 Gy combined with capecitabine 825 mg/m2 bd on radiotherapy days). Patients with a tumor size ≥ 2.5 cm will first undergo concurrent chemoradiotherapy (25x1.8 Gy combined with capecitabine 825 mg/m2 bd on radiotherapy days) to first shrink the tumor and will receive the endoluminal HDR contact boost afterwards in order to eventually fit the tumor surface in the surface of the Maastro applicator.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age and capable of giving informed consent.
* Adenocarcinoma of the rectum classified cT (clinical Tumor) 2-3b, < 5 cm largest diameter and < ½ circumference (MRI staging), N0-N1 (any node < 8 mm diameter), M0
* Operable patient
* Tumor accessible to the Maastro applicator with a distance from the lower tumor border to the anal verge ≤10 cm
* No comorbidity preventing treatment
* Adequate birth control for women of child-bearing potential
* Follow-up possible.

Exclusion Criteria:

* Tumor extending into the anal canal.
* Stop of anti-coagulants (except ≤100 mg aspirin/day) is medically contraindicated.
* Presence of coagulation disorder resulting in an increased bleeding risk.
* Prior pelvic radiation therapy (excluding the abovementioned neoadjuvant treatment).
* Prior surgery or chemotherapy for rectal cancer (excluding the abovementioned neoadjuvant treatment).
* Inflammatory bowel disease (IBD).
* (Systemic) treatment possibly causing rectal or genitourinary toxicity for a separate active malignancy.
* World Health Organization performance status (WHO-PS) ≥ 3.
* Life expectancy of < 6 months.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Clinical feasibility of the Maastro boosting technique. | During treatment
  If at least 7 out of 10 planned Maastro applicator treatment series (3 fractions per series) can be conducted successfully from a procedural point of view the treatment will be considered feasible.

SECONDARY OUTCOMES:
Efficacy of Maastro applicator endoluminal HDR contact brachytherapy boosting in functional organ sparing of the rectum | 3 years follow-up
  Percentage of patients with a persistent clinical complete response with good rectal function (no irreversible G2 or higher toxicity that does not respond to treatment) at 3 years.
  (number of patients with a complete response AND no persistent G2 or higher rectal toxicity) / (total number of patients) * 100%
Percentage of planned interventional Maastro procedures that could be conducted successfully from a procedural point of view. | During treatment
  (procedures conducted successfully from a procedural point of view according to the checklist, please refer to appendix A) / (total number of procedures) * 100%
Duration of the application procedure. | During treatment
  Time from insertion of the proctoscope to finalising removal of the proctoscope in minutes.
Percentage of patients with G3 or higher rectal toxicity up to 3 months after treatment potentially attributable to endoluminal HDR contact brachytherapy. | 3 months follow-up
  Doctor reported CTCEA (Common Terminology Criteria for Adverse Events) v. 5 G3 or higher rectal toxicity not present before the start of treatment and occurring up to 3 months after treatment potentially attributable to endoluminal radiotherapy.
  (number of patients with new G3 or higher rectal toxicity up to 3 months after treatment) / (total number of patients) * 100%
Clinical complete response rate up to 3 years after treatment. | 3 years follow-up
  Clinical response will be assessed using the "watch and wait" protocol which is part of standard clinical care at MUMC+ ( Maastricht Medical University Center). Data will be reported at 3 months, 6 months, 1 year, 2 years and 3 years of follow-up.
  (number of patients with a cCR) / (total number of patients) * 100%
Rectal toxicity scored according to CTCAE v. 5 up to 3 years after treatment. | 3 years follow-up
  Both patient and doctor reported rectal toxicity scored according to CTCEA v. 5 will be determined before each application procedure, weekly during chemoradiotherapy, 1 week after treatment and 1, 3, 6, 12, 18, 24 and 36 months after treatment.
Genitourinary toxicity scored according CTCAE v. 5 up to 3 years after treatment. | 3 years follow-up
  Both patient and doctor reported genitourinary toxicity scored according to CTCEA v. 5 will be determined before each application procedure, weekly during chemoradiotherapy, 1 week after treatment and 1, 3, 6, 12, 18, 24 and 36 months after treatment.
Health status and quality of life as measured by QLQ (quality of life questionnaire)-C30 up to 3 years after treatment. | 3 years follow-up
  Patients will fill out the validated health status and quality of life questionnaire QLQ-C30 after inclusion (at baseline) and 1, 3, 6, 12, 18, 24 and 36 months after treatment.
Health status and quality of life as measured by QLQ-CR29 (Colo Rectal) up to 3 years after treatment. | 3 years follow-up
  Patients will fill out the validated health status and quality of life questionnaire QLQ-CR29 after inclusion (at baseline) and 1, 3, 6, 12, 18, 24 and 36 months after treatment.
Health status and quality of life as measured by EQ-5D (EuroQol Five Dimensions Health Questionnaire) up to 3 years after treatment. | 3 years follow-up
  Patients will fill out the EQ-5D-5L after inclusion (at baseline) and 1, 3, 6, 12, 18, 24 and 36 months after treatment.
Long-term rectal functional outcome as measured by LARS 9 Low Anterior Resection Syndrome) score up to 3 years after treatment. | 3 years follow-up
  Patients will fill out the LARS questionnaire after inclusion (at baseline) and 1, 3, 6, 12, 18, 24 and 36 months after treatment.
Local recurrence rate up to 5 years after treatment. | 5 years follow-up
  Local recurrence rate is defined as the rate of rectal recurrences at the site of the initial primary tumor. Local recurrence rate will be registered up to 5 years after treatment by consulting the hospital patient file.
  (number of patients with a local recurrence) / (total number of patients) * 100%
Locoregional recurrence rate up to 5 years after treatment. | 5 years follow-up
  Locoregional recurrence rate is defined as the rate of recurrences in the rectum and the regional pelvic lymph node areas. Locoregional recurrence rate will be registered up to 5 years after treatment by consulting the hospital patient file.
  (number of patients with a locoregional recurrence) / (total number of patients) * 100%
Metastatic rate up to 5 years after treatment. | 5 years follow-up
  Metastatic rate is defined as the rate of distant metastasis. Metastatic rate will be registered up to 5 years after treatment by consulting the hospital patient file.
  (number of patients with distant metastases) / (total number of patients) * 100%
Salvage surgery rate after treatment. | 5 years follow-up
  The percentage of patients undergoing salvage surgery will be determined. Both TME and local excision rate will be reported separately and combined. The reason for surgery (e.g. local recurrence, patient's wish, unacceptable toxicity) if available and the pathologic outcome (e.g. pCR) will also be reported for patients undergoing surgery. Salvage surgery rate will be registered up to 5 years after treatment by consulting the hospital patient file.
  (number of patients undergoing salvage surgery) / (total number of patients) * 100%
Overall and disease specific survival rate up to 5 year after treatment. | 5 years follow-up
  Both overall survival rate and disease specific survival rates will be reported. Survival rate will be registered up to 5 years after treatment by consulting the hospital patient file.
  100% - (number of patients having died within 5 years after treatment [due to any causes or due to rectal cancer] / total number of patients * 100%)
The diagnostic value of clinical response assessment using digital rectal examination, endoscopy and MRI after endoluminal radiation boosting using the Maastro applicator. | during follow-up
  Clinical response will be assessed using the "watch and wait" protocol which is part of standard clinical care at MUMC+. According to this protocol tumor response is assessed using a digital rectal examination, sigmoidoscopy and MRI (including T2 and DWI). This combined modality approach has been reported to have a specificity of 97% and a sensitivity of 71% for the detection of complete tumor response after neoadjuvant (chemo)radiotherapy. The exact diagnostic value of this multimodality approach has not been validated in the setting of an endoluminal boost with the Maastro applicator. We will evaluate the diagnostic value by relating the test results to a persistent clinical complete response at 1 and 2 years, residual tumor (yes/no) in the resection specimen in case of salvage surgery and a clinical local recurrence in case of refusal of salvage surgery.
Complications within the first 30 days after completion of salvage total mesorectal excision (TME) surgery up to 3 years after treatment. | 3 years follow-up
  Complications within the first 30 days after completion or salvage TME surgery will be scored according to the classification of surgical complications by Clavien-Dindo (16). Complications will be registered up to 3 years after treatment by consulting the hospital patient file.

OTHER OUTCOMES:
Collecting 3D ultrasound measurements of the gross tumor volume (GTV) and intestinal wall layers at every fraction of Maastro applicator brachytherapy. | During treatment
  These images can later be used for scientific research including (but not limited to):
  * Developing a method for ultrasound guided GTV / organs at risk (OAR) (various intestinal wall layers, neighboring organs) dose reconstruction calculation in rectal cancer. This information is crucial in order to establish adequate dose-response relations for tumor control (Tumor Control Probability; TCP) and normal tissue toxicity (Normal Tissue Complication Probability, NTCP). Insight in the dose-response relations will allow the clinician to understand in which way the treatment to the individual patient should be adapted to increase cure rates and/or minimise additional toxicity.
  * Developing ultrasound guided treatment planning software (TPS) which allows future individualised treatment planning.

CONTACTS AND LOCATIONS:
Overall Officials: Maaike Berbée, MD, PhD, Principal Investigator — Maastro, the Netherlands
Locations (1):
- Maastro, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellezzo M, Fonseca GP, Verrijssen AS, Voncken R, Van den Bosch MR, Yoriyaz H, Reniers B, Berbee M, Van Limbergen EJ, Verhaegen F. A novel rectal applicator for contact radiotherapy with HDR 192Ir sources. Brachytherapy. 2018 Nov-Dec;17(6):1037-1044. doi: 10.1016/j.brachy.2018.07.012. Epub 2018 Aug 16. PMID 30122346
- [Background] Bellezzo M, Fonseca GP, Voncken R, Verrijssen AS, Van Beveren C, Roelofs E, Yoriyaz H, Reniers B, Van Limbergen EJ, Berbee M, Verhaegen F. Advanced design, simulation, and dosimetry of a novel rectal applicator for contact brachytherapy with a conventional HDR 192Ir source. Brachytherapy. 2020 Jul-Aug;19(4):544-553. doi: 10.1016/j.brachy.2020.03.009. Epub 2020 May 6. PMID 32386884
- [Background] Gerard JP, Barbet N, Schiappa R, Magne N, Martel I, Mineur L, Deberne M, Zilli T, Dhadda A, Myint AS; ICONE group. Neoadjuvant chemoradiotherapy with radiation dose escalation with contact x-ray brachytherapy boost or external beam radiotherapy boost for organ preservation in early cT2-cT3 rectal adenocarcinoma (OPERA): a phase 3, randomised controlled trial. Lancet Gastroenterol Hepatol. 2023 Apr;8(4):356-367. doi: 10.1016/S2468-1253(22)00392-2. Epub 2023 Feb 16. PMID 36801007